CLINICAL TRIAL: NCT03793634
Title: Evaluation of Topical Chamomile Versus Topical Triamcinolone Acetonide in Management of Oral Lichen Planus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Nashat, 11 saraya st - manial - cairo, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chamomile in OLP
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Chamomile extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The supervisor(AA) will be blind. The principle investigator(EN) will supply the patient with the treatment.
  The supervisor (AA) will assess the clinical parameters before treatment , between visits and at the end of the treatment.
  Statistician will be blind. Double - blind study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- topical chamomile (Experimental): herbal medication which has antioxidant, anti-inflammatory and anticarcinogenesis effect.
  Interventions: Drug: topical chamomile
- Topical Triamcinolone Acetonide (Active Comparator): topical triamcinolone acetonide is the gold standard treatment of oral lichen planus.
  Interventions: Drug: topical chamomile

INTERVENTIONS:
Drug: topical chamomile — herbal medication which has antioxidant, anti-inflammatory and anticarcinogenesis effect

SUMMARY:
Using of herbal medications as topical chamomile which has antioxidant, anti-inflammatory and anticarcinogenesis effect with little side effects is the aim for the future treatment of OLP.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) is a chronic inflammatory T cell mediated autoimmune disease that affects skin and any mucous membrane particularly oral mucosa.The patient complains of burning sensation, pain; interference with eating, swallowing and speech leading to worsening of quality of life.Oxidative stress plays a role in pathomechanism of OLP disease. Enzymatic and non- enzymatic anti-oxidants act as a physiological guard against reactive oxygen species (ROS) and cytokine-mediated toxicity.Herbal treatment is the aim of the future therapy.Chamomile has anti-oxidant , anti-inflammatory effect and accelerate healing.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic OLP.
* Patients with no history of taking corticosteroids for the last 6 months.
* Patients who agree to take medication.
* Medically free

Exclusion Criteria:

* Patients with oral lesions other than OLP.
* Lichenoid reaction .
* Pregnant females and lactation.
* Smokers

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain using Numerical rating scale | 1 month
  Pain measure using Numerical rating scale

SECONDARY OUTCOMES:
clinical sign score | 1 month
  Reduction in clinical sign score using Thongprasom et al